CLINICAL TRIAL: NCT00699790
Title: A 12-Week Randomized, Double-Blinded Study to Evaluate the Effects of Daily Oral Doses of BMS-741672 in Drug-Naive Type 2 Diabetic Patients
Brief Title: Proof of Confidence Study of CCR2 Antagonist (BMS-741672) in Insulin Resistance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB114-005
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; NOS
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: CCR2 Antagonist
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CCR2 Antagonist — Tablets, Oral, 50 mg, once daily, 12 weeks
  Other Names: BMS-741672
  Arms: A1
Drug: Placebo — Tablets, Oral, 0mg, once daily, 12 weeks
  Arms: A2

SUMMARY:
The purpose of the study is to determine whether a CCR2 antagonist (BMS-741672) improves glucose homeostasis in drug-naive type 2 diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* Drug-naive Type 2 diabetics with a screening HbA1c of ≥ 7.5% and ≤ 10%
* Screening FPG ≥ 140 mg/dL and ≤ 220 mg/dL
* BMI ≤ 40 kg/m2

Exclusion Criteria:

* Active tuberculosis
* Symptoms of poorly controlled diabetes
* History of diabetic ketoacidosis
* Significant cardiovascular history or gastrointestinal disorders
* History of unstable or rapidly progressing renal disease
* Active liver disease and/or significant abnormal liver function
* Abnormal chest x-ray at screening indicative of tuberculosis or other infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | after 12 weeks of treatment

SECONDARY OUTCOMES:
Other glycemic, atherosclerosis, lipid and mechanism-based biomarkers will be measured | throughout the 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- Russia (7):
  - Local Institution, Dzerzhnsky
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Saint Petersburg
  - Local Institution, Tyumen
  - Local Institution, Voronezh
  - Local Institution, Yaroslavl

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx